CLINICAL TRIAL: NCT04205474
Title: Aortic Valve Dynamics During Exercise After Valve Sparing Root Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HCH_VSRR_1
Record Dates: First submitted 2019-12-15; First posted 2019-12-19 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Aneurysm Aortic Root; Aortic Valve, Bicuspid
Keywords: valve sparing procedure; reimplantation
MeSH Terms: conditions — Aortic Root Aneurysm; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VSRR with tricuspid aortic valve (Active Comparator): Patients with a tricuspid valve that previously underwent a valve sparing root procedure for aortic root aneurysm
  Interventions: Diagnostic Test: graded bicycle test
- VSRR with bicuspid aortic valve (Active Comparator): Patients with a bicuspid valve that previously underwent a valve sparing root procedure for aortic root aneurysm
  Interventions: Diagnostic Test: graded bicycle test

INTERVENTIONS:
Diagnostic Test: graded bicycle test — the subjects perform an exercise test on a reclining bicycle, and perform against increasing afterload

SUMMARY:
Aortic valve sparing operations are applied in patients with a non-calcified tricuspid or bicuspid aortic valve associated with a root aneurysm, in order to preserve the valve, and avoid new aortic dilatation by stabilizing the aortic valve anulus with a graft prosthesis.

This results in a normal functioning aortic valve, with a low forward gradient across the left ventricular outflow tract.

Little is known about how the repaired aortic valve behaves in conditions of controlled exercise, and how the gradients across the valve change during exercise.

DETAILED DESCRIPTION:
In a cohort of patients operated on since 2000 with a valve sparing operation for aortic root aneurysm in the Department of Cardiac surgery of the University Hospital Ghent, Belgium, and with gradients at rest across the aortic valve of <20mmHg, a graded exercise test on a bicycle (stepwise increase of afterload) will be performed, and the gradient across the aortic valve will be monitored by transthoracic echocardiography at each exercise level. Patients with tricuspid and bicuspid valves will be compared. An age matched, unoperated, and asymptomatic control group with normal functioning tricuspid and bicuspid valves will be examined with the same exercise protocol.

The purpose of the study is the description of the gradients across the aortic valve during exercise, and the discrimination of risk factors that may induce increased gradients.

The hypothesis is that patients with bicuspid valves will demonstrate higher gradients than patients with tricuspid valves, in operated and unoperated individuals.

ELIGIBILITY:
Inclusion Criteria:

* been operated with a valve sparing root procedure in the University Hospital Ghent, Belgium, since 2000
* being able to perform an exercise test on a reclining bicycle
* normal left ventricular function

Exclusion Criteria:

* <18 years or >60 years of age
* peak gradient across the aortic valve at rest of >20mmHg
* decreased left ventricular function

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Echocardiographic gradients in mmHg and velocity across the aortic valve in m/sec at each exercise level | from 1 year postoperatively
  obtained with transthoracic echocardiography during exercise- echocardiographic flow velocity across the aortic valve (colour flow Doppler) and in the left ventricular outflow tract (pulsed-wave Doppler) were measured at regular time intervals during grade exercise, and during recovery - examination was recorded digitally
comparison between peak gradients in mmHg across tricuspid and bicuspid aortic valves | from 1 year postoperatively
  obtained with transthoracic echocardiography during exercise, at each exercise level

SECONDARY OUTCOMES:
comparison between gradients across aortic valve in unoperated and operated patients | 1 year
  gradients in mmHg across the aortic valve, measured by transthoracic echocardiography, at increasing afterload levels, on a reclining bicycle

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Francois, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (1):
- Department of Cardiac Surgery, University Hospital, Ghent, België, Belgium

IPD SHARING:
Plan to Share IPD: No